CLINICAL TRIAL: NCT06018142
Title: Clinical Application of Super-resolution Ultrasound(SR-US) Imaging in Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chief physician, Chinese PLA General Hospital
Other Study IDs: S2023-408-01
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-02

CONDITIONS: Neoplasms, Liver; Neoplasms Malignant; Neoplasm Metastasis; Ultrasound; Microvessels
Keywords: super-resolution ultrasound imaging; ultrasound; solid tumor; micro flow imaging; Microvessels
MeSH Terms: conditions — Liver Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has well accepted that tumor angiogenesis present aberrant vascular architecture and functional abnormalities, which is associated with tumorigenesis, tumor propagation and progression. By locating, separating and tracking microbubbles, the recently introduced and upgraded Ultrasound Localization Microscopy (ULM) surpassed classical wave diffraction limit. However, the acquisition of structural and functional parameters of microcirculation in vivo for ULM is still confined by the compromise between the resolution and penetration depth. The relatively long acquisition time induced the difficulty of motion correction potentially, which hampers the preclinical to clinical application in organs with distinct tissue motion such as the liver. Therefore, we take the lead in studying human liver lesion microvasculature, which remains a challenge for noninvasive, quantitative and functional intravital imaging especially due to its deep-seated location and strong motion. We developed a Super-resolution Ultrasound (SR-US) imaging technique based on ULM to assess its feasibility of visualizing and quantifying microvasculature in human organs.

DETAILED DESCRIPTION:
In this study, 7 indexes were obtained by ultrasonic acquisition. These 7 indicators are used to describe and evaluate the microvessels in the tumor, so as to achieve the early identification and diagnosis of the tumor, and to monitor the growth of the tumor for a long time and evaluate the treatment of the tumor. This is not available with other ultrasound devices.

Based on contrast-enhanced ultrasound, this technology can provide information of smaller blood vessels, which will certainly contribute to the early diagnosis and real-time evaluation of solid tumors during treatment, and play an important role in clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old, gender unlimited;
2. Patients with solid organ tumors with a maximum diameter > 1cm;
3. No contraindications with contrast ultrasound agents;
4. It can improve the pathological results of the tumor or the diagnostic results supported by other relevant imaging tests.
5. Patients can understand the purpose of the examination, voluntarily participate and sign the informed consent.

Exclusion Criteria:

1. The subject is known to be allergic to any component of the contrast agent Sonovue;
2. Lesions were diffuse or borderless on contrast ultrasound;
3. Patients who underwent previous anti-angiogenesis and chemotherapy, or other local treatment of the tumor;
4. Poor image display or deep position in conventional ultrasound evaluation (<10 cm from skin),
5. The researchers determined that there were any other factors that were not suitable for inclusion or affected participants' participation in the study
6. Patients with severe heart disease or lung disease;
7. Patients who are pregnant, may be pregnant or breastfeeding;
8. No enhanced MRI or enhanced CT results can be obtained;
9. The investigator considers the subjects unfit to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for the inclusion criteria as well as the exclusion criteria are enrolled in this study to obtain their clinical information.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Perfusion index | 30 minutes
  The product of the average speed of microbubbles in region of interest (ROI) and the ROI area
Vessel diameter | 30 minutes
  To describe the diameters of the tiniest blood vessels that can be explored
Vessel density | 30 minutes
  To describe the ratio of the number of blood vessels in the tumor to the cross-sectional area of the tumor
Vessel density ratio | 30 minutes
  The ratio of blood vessel density between the core and peripheral areas of the tumor
Mean flow velocity | 30 minutes
  The average velocity in the region of interest
Distance metric | 30 minutes
  The ratio of the total length of the curve path to the straight line distance from the beginning to the end of the curve
Perfusion ratio | 30 minutes
  Perfusion ratio of tumor core to peripheral area

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Department of Interventional Ultrasound of Chinese PLAGH, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The reason we cannot provide individual participant data (IPD) is because the data we obtained from the super-resolution ultrasound images is not publicly available

REFERENCES:
- [Derived] Liang M, Liu J, Wang H, An S, Chen C, Chu H, Zhu M, Su X, Liang P, Zong Y, Wan M. Ultrasound super-resolved hemodynamic estimation in microvessel using physics-informed neural networks and data assimilation. Comput Methods Programs Biomed. 2026 Feb 1;274:109136. doi: 10.1016/j.cmpb.2025.109136. Epub 2025 Oct 30. PMID 41202508
- [Derived] Zeng QQ, An SZ, Chen CN, Wang Z, Liu JC, Wan MX, Zong YJ, Jian XH, Yu J, Liang P. Focal liver lesions: multiparametric microvasculature characterization via super-resolution ultrasound imaging. Eur Radiol Exp. 2024 Dec 5;8(1):138. doi: 10.1186/s41747-024-00540-3. PMID 39636384